CLINICAL TRIAL: NCT05412823
Title: Post Intubation Neurologic Outcomes in Critically Ill Adults
Brief Title: Neurologic Function Post Intubation
Acronym: NeuroHypoxia
Status: Recruiting | Type: Observational
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Dr. Abdullah Bakhsh, Assistant Professor of Emergency Medicine, King Abdulaziz University
Other Study IDs: KAUJED
Record Dates: First submitted 2022-06-05; First posted 2022-06-09 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Intubation Complication
Keywords: Emergency Intubation; Hypoxia; Neurologic Function
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypoxic group: Participants with hypoxia during intubation (after induction and before endotracheal tube placement)
- Non-hypoxic group: Participants without hypoxia during intubation (after induction and before endotracheal tube placement)

SUMMARY:
The frequency of oxygen desaturation during emergency intubation is not uncommon. However, the significance and clinical sequalae of hypoxia during emergency intubation in critically ill, non-trauma patients is not known. Therefore, the aim of this study is to evaluate neurologic function post-intubation of critically ill, non-trauma patients. Providing knowledge on whether the degree of hypoxia during emergency intubation is associated with worse neurologic outcomes, will guide clinical practice to ameliorate that level of hypoxia

DETAILED DESCRIPTION:
Critically ill patients undergoing emergent endotracheal intubation are at risk for oxygen desaturation in a variety of acute care settings. Such complication could arise from patient, operator, or procedure related factors. Evidence suggests that rapid sequence intubation (RSI) improves first-pass success and reduces complications in the critically ill. Nonetheless, the procedure is not without risks. In fact, emergency intubation is associated a reported oxygen desaturation rate of 10.9% - 33.5%. High quality pre-oxygenation has been shown to prolong time to desaturation during emergency airway management. Despite advances preoxygenation techniques, a significant number of patients undergoing emergency intubation still experience desaturation. Most of the time this is transient and easily reversible. Occasionally however, desaturation becomes critical and may result in devastating complications such as dysrhythmias or cardiopulmonary arrest.

The brain consumes a significant amount of energy and is exquisitely sensitive to hypoxia and hypoperfusion. Hypoxic brain injury occurs whenever oxygen delivery to the brain is compromised. The role of secondary brain insults including hypoxia and hypotension, in traumatic brain injury (TBI) is well established. Previous literature has demonstrated that a single event of hypoxemia in a head-injured patient substantially increases morbidity and mortality. This has resulted in airway management being a cornerstone in the care of unconscious TBI patients, to ensure adequate oxygen delivery to the injured brain. However, the significance and clinical sequalae of hypoxia during emergency intubation in critically ill, non-trauma patients is not known. Therefore, the aim of this study is to evaluate neurologic function post-intubation of critically ill, non-trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Good baseline neurologic function (Modified Rankin Scale: 1-3)
* Emergency departments
* Critical care units
* In-patient floors
* Patients undergoing emergent intubations as determined by the treating physician
* Age> 17 years old
* Good baseline modified rankin scale (mRs 1-3)

Exclusion Criteria:

* Pediatric patients (17 years of age of less)
* Pregnant patients
* Intubations occurring in the operating room
* Prisoners
* Trauma
* Status epilepticus
* Primary intracranial pathology
* Cardiopulmonary arrest
* Poor baseline neurologic function (Modified Rankin Scale: 4-5)
* Pre-Hospital Intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adults requiring emergency intubation based on the treating clinician
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRs) | Up to 30-days of intubation
  A validated 6-point scale for measuring the degree of disability in the daily activities of people suffering neurological impairment. The scale runs from 0-6, in which "0" indicates perfect health without disability and "6" indicates the worst outcome which is death.

SECONDARY OUTCOMES:
In-hospital Mortality | Up to 30-days of intubation
  Death during hospital stay
ICU Length of Stay | Up to 30-days from intubation
  Duration of stay in intensive care unit
Hospital Length of Stay | Up to 30-days of intubation
  Duration of stay in hospital
Incidence of Aspiration | Up to 14-days of intubation
  Pulmonary aspiration confirmed by chest X-ray or chest CT
Post-Intubation Complications | Within 24-hours
  Complications arising during the early post-intubation phase

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bodily JB, Webb HR, Weiss SJ, Braude DA. Incidence and Duration of Continuously Measured Oxygen Desaturation During Emergency Department Intubation. Ann Emerg Med. 2016 Mar;67(3):389-95. doi: 10.1016/j.annemergmed.2015.06.006. Epub 2015 Jul 9. PMID 26164643
- [Background] Gebremedhn EG, Mesele D, Aemero D, Alemu E. The incidence of oxygen desaturation during rapid sequence induction and intubation. World J Emerg Med. 2014;5(4):279-85. doi: 10.5847/wjem.j.issn.1920-8642.2014.04.007. PMID 25548602
- [Background] Okubo M, Gibo K, Hagiwara Y, Nakayama Y, Hasegawa K; Japanese Emergency Medicine Network Investigators. The effectiveness of rapid sequence intubation (RSI) versus non-RSI in emergency department: an analysis of multicenter prospective observational study. Int J Emerg Med. 2017 Dec;10(1):1. doi: 10.1186/s12245-017-0129-8. Epub 2017 Jan 25. PMID 28124199
- [Background] Tan E, Loubani O, Kureshi N, Green RS. Does apneic oxygenation prevent desaturation during emergency airway management? A systematic review and meta-analysis. Can J Anaesth. 2018 Aug;65(8):936-949. doi: 10.1007/s12630-018-1124-0. Epub 2018 Apr 23. PMID 29687359
- [Background] Pourmand A, Robinson C, Dorwart K, O'Connell F. Pre-oxygenation: Implications in emergency airway management. Am J Emerg Med. 2017 Aug;35(8):1177-1183. doi: 10.1016/j.ajem.2017.06.006. Epub 2017 Jun 8. PMID 28623005
- [Background] Lacerte M, Hays Shapshak A, Mesfin FB. Hypoxic Brain Injury. 2023 Jan 27. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537310/ PMID 30725995
- [Background] Chesnut RM, Marshall LF, Klauber MR, Blunt BA, Baldwin N, Eisenberg HM, Jane JA, Marmarou A, Foulkes MA. The role of secondary brain injury in determining outcome from severe head injury. J Trauma. 1993 Feb;34(2):216-22. doi: 10.1097/00005373-199302000-00006. PMID 8459458